CLINICAL TRIAL: NCT02712671
Title: Study of Systematic Tuberculosis Testing for Active, Sub-clinical and Latent Tuberculosis Infection in a United Kingdom Human Immunodeficiency Virus (HIV) Infected Cohort
Brief Title: Testing for Tuberculosis in the United Kingdom HIV Infected Population
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Other Study IDs: UCL 12/0212
Record Dates: First submitted 2016-02-29; First posted 2016-03-18 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: HIV; Latent Tuberculosis
Keywords: Cost-Benefit Analysis; Quality of Life
MeSH Terms: conditions — Latent Tuberculosis | interventions — X-Rays; Culture Techniques; Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood plasma and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Enrolled subjects: Subjects attending the Ian Charleson Centre and agreeing to be tested for latent, subclinical and active tuberculosis using Chest radiograph, Blood interferon gamma release assay, Tuberculin skin testing, Sputum induction for mycobacterial microscopy and culture with spirometry, and Mycobacterium tuberculosis polymerase chain reaction testing.
  Interventions: Radiation: Chest radiograph; Procedure: Blood interferon gamma release assay; Procedure: Tuberculin skin testing (TST); Procedure: Sputum induction for mycobacterial microscopy and culture; Other: Mycobacterium tuberculosis polymerase chain reaction testing; Procedure: Spirometry

INTERVENTIONS:
Radiation: Chest radiograph — A chest radiograph involves the participant standing in front of a film and a low dose of radiation passes through the chest. This will be used to look for evidence of tuberculosis infection.
  Other Names: Chest X ray
Procedure: Blood interferon gamma release assay — Test of T-lymphocytes' response to exposure with tuberculosis antigens. This test is used for the diagnosis of latent tuberculosis infection and involves a blood sample in lithium heparin tube. It will be performed in an off site laboratory (Oxford Immunotec, Abingdon, Oxfordshire, United Kingdom).
  Other Names: Blood IGRA; TSpot.TB
Procedure: Tuberculin skin testing (TST) — An intradermal test for latent tuberculosis infection that involves a small injection of purified protein derivative (PPD) from inactivated Mycobacterium tuberculosis. The reaction is interpreted at 48-72 hours by measuring the induration produced.
  Other Names: TST; Mantoux test
Procedure: Sputum induction for mycobacterial microscopy and culture — Participants will breathe in a nebuliser salt solution (3.5% normal saline) for 15 minutes and asked to cough up a sputum sample. This is undertaken in a negative pressure tent. The sample will be tested for mycobacteria under the microscope and then cultured for 42 days in liquid culture bottles the microbiology laboratory.
Other: Mycobacterium tuberculosis polymerase chain reaction testing — Sputum from sputum induction will be tested using the GeneXpert system using polymerase chain reaction to identify genes present in Mycobacterium tuberculosis. This test is performed in a microbiology laboratory and tests for the presence of Mycobacterium tuberculosis in sputum, plus genes associated with drug resistance.
  Other Names: TB PCR; GeneXpert MTB/RIF
Procedure: Spirometry — Participants will be asked to blow into a spirometer to measure how much air they can expel in one second and in a whole breath. This will be repeated six times (three times before inhaling 3.5% saline solution and three times five minutes after breathing 3.5% saline solution). The results will be used to identify those whose airways are sensitive to the solution and to look for the presence of airways disease (asthma or chronic obstructive pulmonary disease).
  Other Names: Lung function

SUMMARY:
Human Immunodeficiency Virus (HIV) is the strongest individual risk factor for the reactivation of tuberculosis (TB) after previous exposure to Mycobacterium tuberculosis (MTb). This risk is reduced but not completely eliminated when HIV is treated with antiretroviral therapy (ART). Both the British HIV Association (BHIVA) and National Institute of Health and Care Excellence (NICE) suggest testing for latent TB infection in HIV infected individuals, but use different criteria. The cost -effectiveness of either approach has not been assessed, nor is testing widespread. A certain proportion of HIV infected subjects in Africa have MTb detectable in their sputum despite not having symptoms (such as cough or weight loss), nor changes on a chest x ray. It is unclear if this happens in lower TB prevalence areas such as the United Kingdom (UK). We intend to test a cohort of HIV infected subjects for evidence of latent TB using a tuberculin skin test (TST) and Interferon Gamma Release Assay (IGRA), ask about symptoms (using a standardised questionnaire) and to induce sputum using a saline nebuliser, to detect MTb using microscopy and culture, and newer nucleic acid amplification (genetic) techniques. Some patients, despite being exposed to TB in the past, will not mount a response using an IGRA or TST, which maybe due to an abnormal immune response. This lack of response seems more common in HIV. By investigating the number of patients with positive TST, IGRA, chest X ray and evidence of MTb in their sputum, in the context of place of birth, previous exposure to TB, CD4 count and other medications, we can assess the cost- effectiveness of systematic TB screening and the use anti-TB antibiotics to prevent reactivation of TB. In time, we will be able to answer important questions about the time taken to reactivate TB in individuals with HIV who do or don't take preventative anti-TB medications in the UK.

DETAILED DESCRIPTION:
The investigators would like to assess a cohort of human immunodeficiency virus (HIV) infected individuals at the Ian Charleson Centre, Royal Free Hospital to assess the rates of latent tuberculosis infection (LTBI) using both tuberculin skin test (TST) and interferon gamma release assay (IGRA), systematically investigating for active tuberculosis (TB) with a symptom questionnaire and chest X ray, and test for Mycobacterium tuberculosis (MTb) in their sputum, both coughed up spontaneously where possible and by inducing sputum using a saline nebuliser and testing this using microscopy and culture (the established method for detecting MTb), nucleic acid amplification testing (using Xpert.TB, a new genetic test for TB that decreases the time required for detection) and a novel 16S ribosomal ribonucleic acid (RNA) test, used to look for TB burden.

A cohort of people with HIV infection will be invited to take part in the study. Subjects will have varying place of origin, TB exposure risk, blood cluster of differentiation 4 (CD4) cell count, HIV viral load, exposure to antiretroviral drugs used to treat HIV. All patients with a new diagnosis of HIV will be invited, as will a group of subjects already undergoing HIV care (selected by stratified sampling) in order to recruit 180 subjects originating from sub-Saharan African countries and 120 from lower TB incidence countries (such as the United Kingdom, UK and Western Europe). The study is powered to detect a difference between all forms of TB infection in subjects from sub-Saharan Africa to those from the UK (or other low TB prevalence countries) with 80% power, allowing a 5% type I error.

The participants will be recruited and a questionnaire, X ray, sputum induction, TST and IGRA can be taken in one visit. They will need to return 48--72 hours later to have the TST read on their arm. Those with evidence of LTBI (with positive TST or IGRA) will be invited to TB/HIV clinic and quality of life scores recorded as part of the study.

Research Questions:

1. To determine the feasibility, yield and cost--effectiveness of testing for M. tuberculosis infection in UK HIV infected individuals.
2. To determine the prevalence of subclinical and active TB in a UK HIV infected clinic
3. To determine the sensitivity and specificity of systematic screening questionnaires for detecting cases of active TB outside of high TB prevalence settings
4. To determine concordance between TST and blood IGRA (T-Spot.TB) in latent TB infection
5. To identify risk factors for latent TB infection in the clinic population
6. To determine the underlying frequency of airways disease (using spirometry) and of respiratory symptoms
7. To determine the sensitivity and specificity of 'Xpert MTB/RIF' polymerase chain reaction (PCR) testing of sputum and induced sputum compared to mycobacterial microscopy and culture
8. To compare the Molecular Bacterial Load (MBL) assay, based on 16S rRNA, and other available molecular assays, with Xpert MTB/RIF for detection of Mtb
9. To determine quality of life scores (EQ-5D) for those with HIV infection, with and without latent TB infection and/or undergoing treatment

   On those with evidence of LTBI:
10. To determine uptake of latent TB therapy (6 months isoniazid treatment)
11. To determine cost of latent TB treatment (including screening costs, clinic time)
12. To determine quality of life and rate and severity of adverse events on latent TB treatment
13. To determine rate and time until active TB in those with LTBI on or off antiretroviral therapy (ART) and/or isoniazid prophylaxis

    In all patients (over 20 year follow up):
14. To determine the rate of incident active TB
15. To determine the time until progression to active TB with in patients with abnormal radiographic changes consistent with old tuberculosis exposure or disease

Data will be generated by the Research team and University College London (UCL) Statistics team.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of HIV or established in care in HIV clinic by stratified sampling
* Able to give informed consent

Exclusion Criteria:

* Diagnosis of active TB or undergoing treatment for active or latent TB
* Inability to produce sputum by coughing (e.g. recent rib fracture, chest pain, pneumothorax)
* Pregnancy
* Use of steroids (equivalent to 15mg prednisolone for ≥4 weeks) or any other immunosuppressive drugs (e.g. azathioprine) - relative
* Active solid organ or haematological malignancy (excluding Kaposi's sarcoma)
* Previous hypersensitivity to purified protein derivative (PPD)
* Extensive eczema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending an ambulatory clinic for Human Immunodeficiency Virus (HIV) care in London.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-06; Primary Completion 2016-02 (Actual); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Number of cases of active tuberculosis disease | 1 year
  Number of cases of active TB disease amongst the enrolled subjects, defined by the number of participants with X ray changes consistent with active tuberculosis and/or sputum culture positive for Mycobacterium tuberculosis with symptoms consistent with tuberculosis disease.
Number of cases of subclinical tuberculosis | 1 year
  Number of cases of subclinical tuberculosis amongst the enrolled subjects, defined by the number of participants with sputum culture positive for Mycobacterium tuberculosis, with or without X ray changes consistent with active tuberculosis and without symptoms consistent with tuberculosis disease.
Number of cases latent tuberculosis infection | 1 year
  Number of cases of latent tuberculosis infection amongst the enrolled subjects, defined by the number of participants with with positive tuberculin skin test (TST) and/or interferon gamma release assay (IGRA) (for latent TB infection), but without a history of previous, treated tuberculosis disease and without symptoms, X ray changes consistent with active tuberculosis disease or sputum culture positive for Mycobacterium tuberculosis.

SECONDARY OUTCOMES:
Number with subsequent active TB disease | 20 years
  Number of participants that develop new TB disease after the testing period has taken place
Time to subsequent active TB disease | 20 years
  Time (months) from when testing took place to subsequent active TB disease in those that develop it.
Number of participants with a diagnosis of airways disease in an HIV infected cohort | 2 years
  Number of participants with symptoms of airways disease (asthma or chronic obstructive pulmonary disease) defined as Forced Expiratory Volume in one second divided by the forced vital capacity <0.7 on spirometry and respiratory symptoms.
Quality of life scores for those with HIV infection with or without TB infection. | 2 years
  Quality of life scores using the EuroQol 5 Dimensions (EQ5D) questionnaire for those with HIV infection, with and without latent TB infection and/or undergoing treatment.
Uptake of latent TB preventive treatment in an HIV clinic cohort | 2 years
  Number of participants that agree to take latent tuberculosis preventive therapy in those with a new diagnosis of latent TB infection divided by the number of patients with a new diagnosis of latent tuberculosis infection.
Cost of latent TB preventive treatment in an HIV clinic cohort | 2 years
  The sum of the costs (£ sterling) associated with preventive treatment for latent tuberculosis infection divided by the number of participants with a diagnosis of latent tuberculosis infection, measured from a United Kingdom National Health Service perspective.
Number of adverse events for each participant taking latent TB preventive treatment | 2 years
  Number and type of adverse events whilst taking latent tuberculosis preventive therapy, measured using standardised adverse effects questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Lipman, MD, Principal Investigator — Clinical Senior Lecturer and Consultant Physician
Locations (1):
- Ian Charleson Centre, Royal Free Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No